CLINICAL TRIAL: NCT06769412
Title: Incidence of Retinal Vasculitis Among Patients Receiving Aflibercept 2 mg: A US Real-World Evidence Study Using the IRIS Registry
Brief Title: A Real-World Evidence Study for the Incidence of Retinal Vasculitis (RV) Among Adult Patients Receiving Aflibercept 2 mg in the United States (US)
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VGFTe-OD-2457
Record Dates: First submitted 2024-12-24; First posted 2025-01-10 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Retinal Vasculitis
Keywords: Anti-vascular endothelial growth factor; Aflibercept; Neovascular age-related macular degeneration (nAMD); Diabetic macular edema (DME); Diabetic retinopathy (DR) without macular edema (ME); Diabetic retinopathy (DR) with macular edema (ME)
MeSH Terms: conditions — Retinal Vasculitis; Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aflibercept IVT Cohort: Patients ≥ 18 years who initiated aflibercept 2 mg IVT during the study period
  Interventions: Drug: aflibercept 2 mg

INTERVENTIONS:
Drug: aflibercept 2 mg — No study-specific investigations for this descriptive observational study
  Other Names: Eylea®

SUMMARY:
This study will describe and estimate the incidence of RV events among patients and patient eyes receiving aflibercept intravitreal (IVT) (Eylea® 2mg) therapy in US clinical practice. This study will also use clinical record review to confirm cases of RV first identified using International Classification of Diseases, tenth revision, Clinical Modification (ICD-10-CM) codes and to identify RV with occlusion.

DETAILED DESCRIPTION:
This study is purely descriptive using secondary data from the Verana Health Retinal Outcomes module sourced from the American Academy of Ophthalmology's Intelligent Research in Sight (IRIS®) Registry

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient-eyes with at least one aflibercept 2 mg injection between January 1, 2017 and June 30, 2023
2. Patient-eyes with at least one aflibercept 2 mg injection with a specified laterality. The earliest date of aflibercept injection will be the index date for each patient-eye
3. Patient-eyes with diagnosis (documented through ICD-10-CM diagnosis code) of nAMD, DME, DR without DME, DR with ME status unknown, and/or ME following RVO in the same eye as the aflibercept injection within 14 days prior to the index date (inclusive)

Key Exclusion Criteria:

1. Patients with aflibercept 2 mg injection within 12 months (365 days) prior to the index date (not inclusive) will be excluded, as defined in the protocol
2. Patient-eyes with a diagnosis of RV in the same eye as the aflibercept injection or with unspecified laterality within 12 months (365 days) prior to index date (inclusive), as defined in the protocol
3. Aflibercept treatment episodes (aflibercept injections) with unspecified laterality, ophthalmic procedures or surgeries within 60 days prior to the injection date

NOTE: Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will represent patients and patient-eyes who initiate aflibercept 2 mg injections to treat neovascular age-related macular degeneration (nAMD), diabetic macular edema (DME), diabetic retinopathy (DR) without DME, DR with macular edema (ME) status unknown, or ME following retinal vein occlusion (RVO).
Sampling Method: Non-Probability Sample
Enrollment: 550000 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of RV events | During the 60-Day at-risk period following aflibercept 2 mg IVT, up to approximately 6.5 years
Incidence of occlusive RV events confirmed through clinical chart abstraction | During the 60-Day at-risk period following aflibercept 2 mg IVT, up to approximately 6.5 years
Incidence of non-occlusive RV events confirmed through clinical chart abstraction | During the 60-Day at-risk period following aflibercept 2 mg IVT, up to approximately 6.5 years
Incidence of unconfirmed RV events | During the 60-Day at-risk period following aflibercept 2 mg IVT, up to approximately 6.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Regeneron Research Site, Tarrytown, New York, United States